CLINICAL TRIAL: NCT01101945
Title: An Open Label, Multi-Center, Long-Term Follow-up Study to Evaluate the Safety of PHX1149T in Subjects With Type 2 Diabetes Mellitus - Extension to Protocol PHX1149-PROT202
Brief Title: Long-term Extension Study to Evaluate the Safety of Dutogliptin/PHX1149T in Subjects With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Phenomix (Industry)
Responsible Party: Hans-Peter Guler, MD, Phenomix Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHX1149-PROT202E
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; DPP4 inhibitor; dutogliptin; PHX1149
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dutogliptin

INTERVENTIONS:
Drug: dutogliptin — 400 mg QD

SUMMARY:
The purpose of this study is to demonstrate that dutogliptin/PHX1149T is safe and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Completed Visit 7/Day 98 of the core protocol PHX1149-PROT202
* Current treatment of Type 2 diabetes mellitus in accordance with product labeling with metformin, or thiazolidinedione (TZD), or metformin + TZD

Exclusion Criteria:

* Inadequately controlled Type 2 diabetes mellitus with need for therapy with insulin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
To demonstrate safety and tolerability of dutogliptin/PHX1149T as assessed by vital signs, adverse event reporting, and routine clinical laboratory assessments | 104 weeks
To demonstrate safety and tolerability of dutogliptin/PHX1149Tas assessed by vital signs, adverse event reporting, and routine clinical laboratory assessments | 208 weeks (U.S. only)

SECONDARY OUTCOMES:
To demonstrate maintenance or lowering of HbA1c and fasting blood glucose | 104 weeks

CONTACTS AND LOCATIONS:
Locations (55):
- United States (27):
  - Fullerton, California
  - Long Beach, California
  - Orange, California
  - San Diego, California
  - Kissimmee, Florida
  - Melbourne, Florida
  - New Port Richey, Florida
  - Gurnee, Illinois
  - Wichita, Kansas
  - Kansas City, Missouri
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Berlin, New Jersey
  - Margate City, New Jersey
  - Trenton, New Jersey
  - Charlotte, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Medford, Oregon
  - Warminster, Pennsylvania
  - Columbia, South Carolina
  - Greer, South Carolina
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Norfolk, Virginia
- Argentina (6):
  - Cuidad Autonoma de Buenos Aires, Buenos Aires
  - La Plata, Buenos Aires
  - Lanús Este, Buenos Aires
  - Morón, Buenos Aires
  - Quilmes, Buenos Aires
  - Corrientes, Corrientes Province
- Canada (11):
  - Calgary, Alberta
  - Red Deer, Alberta
  - Mount Pearl, Newfoundland and Labrador
  - St. John's, Newfoundland and Labrador
  - Etobicoke, Ontario
  - London, Ontario
  - Samia, Ontario
  - Toronto, Ontario
  - Cornwall, Prince Edward Island
  - Mirabel, Quebec
  - Montreal, Quebec
- India (7):
  - Ellisbridge, Ahmedabad
  - Banjara Hills, Hyderabad
  - Punjagutta, Hyderabad
  - Pune, Maharashtra
  - Tardeo, Mumbai
  - Dhantoli, Nagpur
  - Chennai, Tamil Nadu
- Mexico (4):
  - Guadalajara, Jalisco
  - Mexico City, Mexico City
  - Morelia, Michoacán
  - Monterrey N. L., Nuevo León